CLINICAL TRIAL: NCT00191256
Title: Randomized Phase II Trial to Outline the Efficacy of Gemcitabine Containing Regimens (Gemcitabine/Carboplatin and Gemcitabine/Paclitaxel) When Used as Preoperative Chemotherapy In Patients With Stage I and II NSCLC
Brief Title: Efficacy Trial of Gemcitabine Containing Regimens As Preoperative Chemotherapy in Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5488; B9E-US-S235
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Carcinoma, Non Small Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Carboplatin; Paclitaxel

INTERVENTIONS:
Drug: Gemcitabine
Drug: Carboplatin
Drug: Paclitaxel

SUMMARY:
To evaluate the rate of complete pathological response after 3 cycles of gemcitabine containing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non small cell lung cancer
* No prior chemotherapy or radiation for non small cell lung cancer
* No prior malignancy

Exclusion Criteria:

* Pregnancy or breastfeeding
* Serious concomitant disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77
Dates: Start 2001-06; Study Completion 2006-07

PRIMARY OUTCOMES:
Pathological complete response rate, in previously untreated patients with clinical Stage I and II non-small cell lung cancer (NSCLC).

SECONDARY OUTCOMES:
Response rate, disease free survival,toxicities including pulmonary toxicity, operative mortality, and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina, United States